CLINICAL TRIAL: NCT02136849
Title: Inter-regional Project of the Great Western Exploration Approach for Exome Molecular Causes Severe Intellectual Disability Isolated or Syndromic
Acronym: HUGODIMS
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Collaborators: Nantes Genomics platform (Unknown)
Responsible Party: Sponsor
Other Study IDs: RC14_0107
Record Dates: First submitted 2014-05-09; First posted 2014-05-13 (Estimated); Last update posted 2018-12-12 (Actual); Status verified 2016-03

CONDITIONS: Severe Intellectual Disability
Keywords: severe intellectual disability, genetic, de novo exome
MeSH Terms: conditions — Intellectual Disability

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 2 tubes of 5 ml EDTA blood
Oversight: Data Monitoring Committee: No

SUMMARY:
Intellectual disability (ID) moderate or severe affects about one child in 250, with 3000 to 4000 new cases each year. Chromosomal or molecular pathology causes are not identified in half of the cases by current techniques. Studies show that de novo mutations are common in many different genes. The "exome" approach by high-throughput sequencing (NGS) has emerged as the technique of choice for identifying and comparing the exome of the child to the parent. We wish to evaluate this approach and its contribution in the diagnostic management of 50 patients with DI seen in genetics in 6 CHU Great West. Genomics platform IBISA / Biogenouest will provide technological and bioinformatics support this project.

ELIGIBILITY:
Inclusion Criteria:

* Patients with severe intellectual disability (IQ <35 ) or moderate (IQ <50) isolated or syndromic presentation but undiagnosed . The diagnosis is established during genetic counseling of a 6 CHU interregion
* Lack of family history ( parents). We are interested in this project to patients who do not have family history in order to increase the probability of identifying a de novo mutation . We do not however exclude the hypothesis for some patients a mechanism recessive autosomal or X-linked .
* Recruitment in 6 CHU HUGO . Patients are required to have been seen in genetics in a 6 CHU interregion . Molecular analyzes of the Fragile X syndrome and the CGH technique must be negative.
* Indication sequencing exomique adopted by the Scientific Committee. The Scientific Committee HUGODIMS project role to select patients whose DNA will be studied in order to optimize the chances of success for sequencing . This selection must take into account clinical parameters , but also genetic parameters ( potential inbreeding ) . The files will be selected by videoconferencing at the end of the monthly meeting of CLAD . The methodologist of the study will be invited to videoconferencing.
* specific consent obtained for the study.

Exclusion Criteria:

* Parents patient with moderate or severe intellectual disability disagree with the preferred hypothesis of de novo mutation or recessive transmission mechanism.
* Form with known syndromic diagnosis can be targeted molecular studies (clinical signs).
* Cause molecular DI identified by targeted molecular analysis or CGH.
* Explicit refusal to participate in the study of the patient, parents, or one of the two parents.
* Any other indication that intellectual disability.
* The parents of the patient or the patient may be removed.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: We planned to include 50 trios (patients + parents) in the study. This number appears to be sufficient to achieve the defined objectives and according to the literature data (Rauch et al, 2012).
  The study population is the population affected by severe intellectual disability according to the commonly accepted definition (IQ <35), and patients with severe or moderate ID (IQ <50) associated with other clinical signs but no obvious syndromic form known . In 2 cases, the parents of patients will not be affected by DI. The recruitment will be made during genetic counseling. Many patients with DI meet the criteria of the study are already being explored in different centers. For these patients, the DNA of the index case and parents is already available. Families will therefore re-contacted to invite them to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 228 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Number of patients for which a mutation responsible for the de novo patients DI has been identified | 18 months

SECONDARY OUTCOMES:
Number of patients for whom the study of exomes revealed mutations in genes compatible with the mode of recessive autosomal recessive or X-linked chromosome | 18 months
Number of de novo mutations (loss of function, missense or indels) probably pathogens identified are not known to be involved in the DI genes. | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane Bézieau, Pr, Principal Investigator — Nantes University Hospital
Locations (5):
- France (5):
  - Angers University Hospital, Angers
  - Brest University Hospital, Brest
  - Poitiers University Hospital, Poitiers
  - Rennes University Hospital, Rennes
  - Tours University Hospital, Tours